CLINICAL TRIAL: NCT07272980
Title: Three-Session Non-Surgical Periodontal Therapy Improves Biochemical and Microbiological Profiles in Patients With Severe Grade C Periodontitis
Acronym: TSTG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gülnur Emingil (Other)
Collaborators: Ege University Scientific Research Projects Coordination Unit (Unknown)
Responsible Party: Sponsor-Investigator, Gülnur Emingil, Principal Investigator, Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-DİŞ-006
Record Dates: First submitted 2025-11-13; First posted 2025-12-09 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-10

CONDITIONS: Periodontitis (Stage 3); Periodontitis Stage III
Keywords: non-surgical periodontal therapy; scaling and root planning; periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Intervention Model Description: Participants with Stage III/IV Grade C periodontitis were randomly assigned to one of two treatment groups: a single-session scaling and root planing (SRP) protocol or a three-session SRP protocol. Both groups received the allocated intervention in parallel and were followed for 6 months. A healthy control group was also included for comparison.
Who Masked: Outcomes Assessor
Masking Description: Single-blinded design: Outcome assessors were blinded to treatment allocation, while participants and care providers were aware of the assigned intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single-session non-surgical periodontal therapy (Experimental): Participants received full-mouth scaling and root planing (SRP) completed in a single session under local anesthesia. Standard oral hygiene instructions were provided.
  Interventions: Procedure: Scaling and Root Planing (SRP)
- Three-session non-surgical periodontal therapy (Experimental): Participants received full-mouth scaling and root planing (SRP) over three consecutive weekly sessions under local anesthesia. Standard oral hygiene instructions were provided.
  Interventions: Procedure: Scaling and Root Planing (SRP)
- Healthy control group (No Intervention): Periodontally healthy participants without clinical attachment loss or probing depths ≥4 mm were examined and sampled but received no periodontal treatment.

INTERVENTIONS:
Procedure: Scaling and Root Planing (SRP) — Full-mouth scaling and root planing (SRP) performed under local anesthesia, either in a single session or divided into three weekly sessions depending on the study arm. Standard oral hygiene instructions were provided to all participants.
  Arms: Single-session non-surgical periodontal therapy; Three-session non-surgical periodontal therapy

SUMMARY:
This clinical study investigates two different non-surgical periodontal therapy approaches in patients with advanced periodontitis and compares them with periodontally healthy individuals. Participants with Stage III/IV Grade C periodontitis are randomly assigned to either a single-session or a three-session scaling and root planing (SRP) protocol. Clinical parameters, gingival crevicular fluid inflammatory markers, and subgingival microbial profiles are assessed at baseline and during a 6-month follow-up period. The study aims to determine whether performing non-surgical periodontal therapy in multiple sessions influences clinical, biochemical, and microbiological responses.

DETAILED DESCRIPTION:
This randomized, single-blinded, controlled clinical trial is conducted at the Department of Periodontology, School of Dentistry, Ege University, İzmir, Turkey. The purpose of the study is to evaluate whether a three-session non-surgical periodontal therapy protocol provides different clinical, biochemical, and microbiological responses compared to a single-session protocol in patients with Stage III/IV Grade C periodontitis.

Participants with periodontitis are randomly assigned to one of two intervention groups:

Single-Session Therapy Group (SSTG): full-mouth scaling and root planing (SRP) performed in one visit.

Three-Session Therapy Group (TSTG): quadrant-wise SRP delivered over three sessions within the same week.

All procedures are carried out by a single calibrated clinician. Clinical periodontal parameters-probing depth, clinical attachment level, plaque index, and bleeding on probing-are recorded at baseline and at predetermined follow-up visits at 1, 3, and 6 months.

Gingival crevicular fluid samples are collected to quantify inflammatory biomarkers, including interleukin-1β (IL-1β), interleukin-6 (IL-6), clusterin, cystatin C, and osteocalcin, using multiplex immunoassays. Subgingival microbial profiles are evaluated using checkerboard DNA-DNA hybridization targeting a panel of selected bacterial species.

The study protocol has received ethics approval from the Ege University School of Medicine Ethics Committee, and written informed consent is obtained from all participants. The research is supported by the Scientific Research Projects Coordination Unit of Ege University.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy, non-smoking individuals aged 18-65 years
* Diagnosis of Stage III or IV Grade C periodontitis according to the 2018 classification of periodontal diseases
* Presence of at least 20 teeth
* No periodontal treatment within the previous 6 months
* Willingness to participate and provide written informed consent

Exclusion Criteria:

* Presence of systemic diseases or conditions affecting the periodontium (e.g., diabetes mellitus, cardiovascular diseases, immunological disorders)
* Pregnancy or lactation
* Use of antibiotics, anti-inflammatory, or immunosuppressive drugs within the past 3 months
* History of periodontal therapy or surgery within the last 6 months
* Smoking or use of any tobacco products

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-11-21 (Actual); Primary Completion 2011-05-22 (Actual); Study Completion 2011-05-22 (Actual)

PRIMARY OUTCOMES:
Change in Full-Mouth Mean Probing Depth (PD) | Baseline to 6 months
  Mean change in probing depth (in millimeters) measured at six sites per tooth from baseline to 6 months.

SECONDARY OUTCOMES:
Change in Clinical Attachment Level (CAL) | Baseline, 1 month, 3 months, and 6 months after treatment
  Evaluation of changes in CAL (mm) at six sites per tooth to assess periodontal healing and inflammation following single-session versus three-session scaling and root planing (SRP).
Change in Bleeding on Probing (BOP) | Baseline, 1 month, 3 months, 6 months
  Change in BOP (%), measured as the percentage of sites exhibiting bleeding on gentle probing, to assess gingival inflammation.
Change in Plaque Index (PI) | Baseline, 1 month, 3 months, 6 months
  Change in PI to evaluate supragingival plaque levels, assessed as the percentage of tooth surfaces with visible supragingival plaque, to evaluate the level of supragingival biofilm accumulation.
Change in Gingival Crevicular Fluid Biomarker Levels (Clusterin, Cystatin C, IL-1β, IL-6, and Osteocalcin) | Baseline, 1 month, 3 months, and 6 months after treatment
  GCF samples collected from sites with PD ≥ 5 mm will be analyzed using multiplex immunoassay to determine changes in host-response biomarkers reflecting tissue inflammation and repair.
Change in Subgingival Microbiota Composition | Baseline, 1 month, 3 months, and 6 months after treatment
  Quantitative and qualitative assessment of periodontal pathogens (e.g., A. actinomycetemcomitans, P. gingivalis, T. denticola, T. forsythia, F. nucleatum) via DNA-DNA checkerboard hybridization to evaluate microbiological effects of SRP regimens.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, School of Dentistry, Istanbul, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) underlying this article will not be shared because anonymized patient-level data were analyzed only in aggregate form, and no separate data repository was created for public access. Summary results are fully presented in the published article.